CLINICAL TRIAL: NCT05122754
Title: Switching From Tenofovir Disoproxil Fumarate-based Antiretroviral Therapy Regimens to Bictegravir/Emtricitabine/Tenofovir Alafenamide in Virally Suppressed Adults With HIV-1 Infection
Brief Title: Switching From TDF-based Antiretroviral Therapy Regimens to B/F/TAF in Virally Suppressed Adults With HIV-1 Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: Xixi Hospital of Hangzhou (Unknown); Yunnan AIDS Care Center (Other)
Responsible Party: Principal Investigator, Jun Chen, MD, Deputy Director of Department of Infectious Diseases and Immunology, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B/F/TAF
Record Dates: First submitted 2021-10-21; First posted 2021-11-17 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: HIV-1-infection
Keywords: Bictegravir/Emtricitabine/Tenofovir alafenamide; Tenofovir Disoproxil Fumarate; HIV-1 infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- B/F/TAF group (Experimental): Bictegravir/emtricitabine/tenofovir alafenamide for 48 weeks.
  Interventions: Drug: B/F/TAF
- TDF-based triple ART regimen switching to B/F/TAF (Active Comparator): TDF-based triple ART regimen for 24 weeks, and all switch to bictegravir/emtricitabine/tenofovir alafenamide for the later 24 weeks.
  Interventions: Drug: TDF-based triple ART regimen switching to B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — Bictegravir/emtricitabine/tenofovir alafenamide once daily, 1 tablet at a time, with or without food for 48 weeks.
  Arms: B/F/TAF group
Drug: TDF-based triple ART regimen switching to B/F/TAF — Tenofovir disoproxil fumarate was administered once daily, one tablet at a time, with or without food. After Week 24, control subjects were also switched to bictegravir/emtricitabine/tenofovir alafenamide once daily, one tablet at a time, with or without food for the later 24 weeks.
  Arms: TDF-based triple ART regimen switching to B/F/TAF

SUMMARY:
To evaluate the safety and efficacy of bictegravir/emtricitabine/tenofovir alafenamide versus tenofovir disoproxil fumarate-based antiretroviral regimens in HIV-infected individuals with virological suppression.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, controlled, open labeled clinical trial, which aims to evaluate the safety and efficacy of B/F/TAF versus TDF-based antiretroviral therapy in HIV-infected individuals with virological suppression, and to evaluate the changes in quality of life and adherence after switching from a TDF-based regimen to B/F/TAF in HIV-infected individuals with virological suppression.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Diagnostic Criteria for AIDS or HIV Infection (WS 293-2019);
* Age 18 or above (included 18);
* Continuous administration of a TDF-based triple ART regimen with a backbone of non-nucleoside reverse transcriptase or protease inhibitors ≥24 weeks and ongoing use;
* Maintaining virological suppression (viral load < 50 copies/mL) for ≥ 24 weeks, and maintaining virological suppression at present;
* Glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73 m2 (calculated according to the CKD-EPI formula);
* ECG is normal;
* White blood cell count ≥3×109/L, Neutrophil count ≥1.5×109/L, Hemoglobin ≥90 g/L, and Platelet count ≥ 75×109/L;
* Alanine aminotransferase and aspartate aminotransferase ≤5×ULN, direct bilirubin ≤1.5×ULN, amylase≤2×ULN；
* Those who volunteered for this study and were able to complete all follow-up visits and sign the informed consent form in accordance with the protocol.

Exclusion Criteria:

* In the 30 days(inclusive) before the screening period, an AIDS-related opportunistic infection or tumor occurred;
* History of known past HIV resistance (confirmed HIV viral load > 200 copies /ml) or resistance to any nucleoside (acid) analogues;
* Decompensated liver cirrhosis;
* Female subject who has a positive urine pregnancy test;
* Lactating women;
* Women who are unable to take a reasonable method of contraception during the trial (including the Screening Period and 30 days after discontinuation of experimental drugs);
* Subjects had other medical conditions requiring treatment with either of the current ART regimens or other drugs which have drug-drug interaction with B/F/TAF and cannot be discontinued.
* Being involved in other interventional clinical studies;
* Those with allergic constitution or known allergy to the components of the drug;
* Suffering from serious mental or neurological diseases;
* Suspected or confirmed history of alcohol and drug abuse; Patients who were not considered by the investigator to be suitable for participating in this clinical trial (such as weak constitution, poor compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in spine and hip bone mineral density (DXA) at 48 weeks | From baseline to Week 48

SECONDARY OUTCOMES:
Percentage change from baseline in spine and hip bone mineral density (DXA) at Week 24 | From baseline to Week 24
The percentage of subjects with spine or hip bone mineral density (DXA) that increased or decreased by more than 3% (not included) from baseline at Weeks 24 and 48 | From baseline to Week 24, 48
Changes from Baseline in Spine and Hip Bone Mineral Density T-Values (DXA) at Weeks 24 and 48 | From baseline to Week 24, 48
Changes from Baseline in eGFR at Weeks 24 and 48 (CKD-EPI Formula) | From baseline to Week 24, 48
The percentage of subjects with HIV viral load < 50 copies /ml at Weeks 24 and 48 | From baseline to Week 24, 48
Changes from baseline in CD4 T cell count at Weeks 24 and 48 | From baseline to Week 24, 48
Changes from baseline in CD4/CD8 ratio at Weeks 24 and 48 | From baseline to Week 24, 48
Changes from baseline in blood lipid (TC, TG, LDL, HDL) at Weeks 24 and 48 | From baseline to Week 24, 48
Quality of life score (WHO QOL-BREF-HIV Scale) change from baseline at Weeks 24 and 48 | From baseline to Week 24, 48
Adherence (Visual Analog Scale) change from baseline at Weeks 24 and 48 | From baseline to Week 24, 48
Patients reported outcome using SSC-HIV-SC scale | From baseline to Week 24, 48

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D, Principal Investigator — Shanghai Public Health Clinical Center
Locations (3):
- China (3):
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Yunnan AIDS Care Center, Kunming, Yunnan
  - Xixi hospital of Hangzhou, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shao Y, Yang X, Yu J, Wang X, Wang J, Liu M, Yang Z, Han J, Zhang R, Liu L, Shen Y, Sun M, Wu L, Zheng Z, Tang Y, Yang J, Wang Z, Qi T, Xu S, Xun J, Sun J, Song W, Chen J. Bone Mineral Density Changes in People with HIV Who had Immediate Switch Versus Deferred Switch from Tenofovir Disoproxil Fumarate-Based Regimens to Bictegravir/Emtricitabine/Tenofovir Alafenamide: A Multicenter, Open-Label, Randomized Clinical Trial. Infect Dis Ther. 2026 Jan;15(1):165-181. doi: 10.1007/s40121-025-01262-8. Epub 2025 Nov 21. PMID 41266678